CLINICAL TRIAL: NCT01446510
Title: Systematic Review and Meta-Analysis of Venous Thromboembolism Risk Assessment Models in Hospitalized Medical Patients
Brief Title: Systematic Review and Meta-Analysis of Venous Thromboembolism (VTE) Risk Assessment in Hospitalized Medical Patients
Status: Withdrawn | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: VTERiskMA8011
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2011-09

CONDITIONS: Venous Thromboembolism
Keywords: VTE; DVT; PE; Risk assessment; risk score; risk analysis; Venous thromboembolism risk
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized Medical Patients: All hospitalized medical adult patients
  Interventions: Other: Application of VTE Risk Assessment

INTERVENTIONS:
Other: Application of VTE Risk Assessment — Use of a method to assess a patient's risk of VTE, and then appropriate prophylaxis for the assigned level of risk

SUMMARY:
A systematic review and meta analysis will be performed of risk assessment models for Venous thromboembolism ("VTE" including pulmonary embolism "PE" and deep venous thrombosis "DVT")in hospitalized medical patients. The goal of this study is to evaluate whether the incidence of VTE is lower in patients that are evaluated with a risk assessment model and treated with thromboprophylaxis for their assigned level of risk.

DETAILED DESCRIPTION:
Venous thromboembolism ("VTE" including pulmonary embolism "PE" and deep venous thrombosis "DVT") is associated with significant morbidity and mortality. Only about half of eligible hospitalized medical patients receive appropriate thromboprophylaxis. Understanding VTE risk factors predictive of VTE among hospitalized medical patients may promote superior thromboprophylaxis. To date a systematic review of VTE risk assessment strategies among hospitalized medical patients, and a meta-analysis reporting the rate of VTE among patient groups at varying levels of risk for VTE does not exist.

The investigators will use the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) checklist for reporting systematic reviews and meta-analyses to develop this systematic review and meta-analysis.

The investigators will perform a systematic review of the literature and report VTE risk assessment models that have been derived and validated among hospitalized medical patients. The investigators will perform a meta-analysis of studies that report a rate of VTE among patients identified as being at elevated risk for VTE and those that are not. The investigators pre-specify that they are going to analyze the prospective and retrospective studies captured by the literature search in two ways. First, the investigators will perform an analysis that groups both prospective and retrospective studies together. The investigators will also perform an analysis that separates out the prospective and retrospective studies. While this will decrease our sample size (and thus power), this approach may allow us to identify any bias or confounding present due to the retrospective study design and then control for it. Notably confirmation that both retrospective and prospective studies identified the same findings would enhance the clinical usefulness of our findings.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Hospitalized

Exclusion Criteria:

* Surgical patients
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized medical patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
VTE | 28 to 180 days
  Objectively confirmed within individual studies

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Woller, MD, Study Director — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

REFERENCES:
- [Background] Liberati A, Altman DG, Tetzlaff J, Mulrow C, Gotzsche PC, Ioannidis JP, Clarke M, Devereaux PJ, Kleijnen J, Moher D. The PRISMA statement for reporting systematic reviews and meta-analyses of studies that evaluate healthcare interventions: explanation and elaboration. BMJ. 2009 Jul 21;339:b2700. doi: 10.1136/bmj.b2700. PMID 19622552
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Quiroz R, Kucher N, Zou KH, Kipfmueller F, Costello P, Goldhaber SZ, Schoepf UJ. Clinical validity of a negative computed tomography scan in patients with suspected pulmonary embolism: a systematic review. JAMA. 2005 Apr 27;293(16):2012-7. doi: 10.1001/jama.293.16.2012. PMID 15855435